CLINICAL TRIAL: NCT02802982
Title: Mathematical Modeling to Predict the Duration of Thrombocytopenia in Neonates
Status: Active, not recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Iowa (Other)
Responsible Party: Principal Investigator, Martha Sola-Visner, MD, Boston Children's Hospital
Other Study IDs: IRB-P00005413; 5R01HL069990-11 (NIH)
Record Dates: First submitted 2016-06-14; First posted 2016-06-16 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Neonatal Thrombocytopenia
Keywords: Thrombocytopenia; Neonates
MeSH Terms: conditions — Thrombocytopenia, Neonatal Alloimmune; Thrombocytopenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A single blood sample drawn (approx. 800 mcL total) for a complete blood count with IPF and for determination of a panel of factors important in the regulation of thrombopoiesis (including TPO, IL-6, IL-11, IL-3, PF-4, VEGF, IGF-1, IGF-II, TGF-ß, HGF, PDGF, and Epo).
  In addition, left-over blood from clinically indicated studies will be collected from the clinical laboratory, processed and stored at -80C for future cytokine studies. Samples will continue to be collected and serial platelet counts with IPF followed until resolution of the thrombocytopenia, defined as a platelet count >60,000/uL for five days without platelet transfusions.
Oversight: Data Monitoring Committee: No

SUMMARY:
Parents of infants who have been thrombocytopenic for 3-4 days will be approached for consent to enter the study. For the purposes of the study, thrombocytopenia will be defined as a platelet count <60,000/uL or a platelet count <100,000/uL that prompted a platelet transfusion. Following enrollment, the platelet count will be followed in each infant. Participants will enter the study if on day 5 or later after the onset of thrombocytopenia (defined as above) infants either have a platelet count <60,000/uL or a platelet count <100,000/uL for which a platelet transfusion is ordered.

DETAILED DESCRIPTION:
Parents of infants who have been thrombocytopenic for 3-4 days will be approached for consent to enter the study. For the purposes of the study, thrombocytopenia will be defined as a platelet count <60,000/uL or a platelet count <100,000/uL that prompted a platelet transfusion. Following enrollment, the platelet count will be followed in each infant. Participants will enter the study if, on day 5 or later after the onset of thrombocytopenia (defined as above), infants either have a platelet count <60,000/uL or a platelet count <100,000/uL for which a platelet transfusion is ordered. If criteria are met, eligible infants will have a single blood sample drawn (approx. 800 mcL total) for a complete blood count with Immature Platelet Fraction (IPF) and for determination of a panel of factors important in the regulation of thrombopoiesis (including TPO, IL-6, IL-11, IL-3, PF-4, VEGF, HGF, PDGF, and Epo). Importantly, in patients who are being transfused for platelet counts <100,000/uL, this sample will need to be obtained immediately prior to the platelet transfusion. If the patient has a platelet count <60,000/uL and is not being transfused, the blood can be obtained at any time.

Following this initial sample, a platelet count with IPF will be obtained any time a CBC is ordered for clinical indications, using left-over blood stored in the clinical laboratory for <24 hrs (only 100 mcL are needed for this). In addition, left-over blood from clinically indicated studies will be collected from the clinical laboratory, processed and stored at -80C for future cytokine studies. Samples will continue to be collected and serial platelet counts with IPF followed until resolution of the thrombocytopenia, defined as a platelet count >60,000/uL for five days without platelet transfusions.

In addition, research nurses will collect and record the infants' demographic data (including gestational age, days of life, birth weight), diagnoses, clinical condition at the time of study entry (respiratory and/or hemodynamic support), time and volume of platelet transfusions, coagulation tests, liver enzymes, and tests of kidney function. Moderate and severe bleeding will also be recorded, using criteria defined a priori.

ELIGIBILITY:
Inclusion Criteria:

1. Are admitted to one of the participating NICUs or the CICU at BCH;
2. Have a post-conceptional age (gestational age + age in weeks) between 23 and 48 weeks; and
3. Have had thrombocytopenia, defined as a platelet count <60,000/uL or a platelet count <100,000/uL but receiving platelet transfusions, for ≥ 5 days.

Exclusion Criteria:

1. Are on ECMO; or
2. Are not expected to survive by the attending neonatologist.

Ages: 5 Days to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants who have been thrombocytopenic for 5 days will be approached for the study.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2013-04; Primary Completion 2016-12 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Prediction of the duration of thrombocytopenia in neonates. | 3 years
  to develop clinically useful parameters to predict the duration of thrombocytopenia in neonates, using mathematical modeling.

CONTACTS AND LOCATIONS:
Overall Officials: Martha Sola-Visner, MD, Principal Investigator — Boston Children's Hospital
Locations (3):
- United States (3):
  - The University of Iowa, Iowa City, Iowa
  - Boston Children's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No